CLINICAL TRIAL: NCT03999411
Title: A Novel Smartphone-based Intervention to Support Smoking Cessation and Adherence to Antiretroviral Therapy Among People Living With HIV: A Pilot Randomized Clinical Trial
Brief Title: Smartphone Intervention for Smoking Cessation and Improving Adherence to Treatment Among HIV Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Taghrid Asfar, Research Assistant Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20190181
Record Dates: First submitted 2019-06-24; First posted 2019-06-26 (Actual); Results first posted 2021-12-02 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Smoking; Smoking Cessation; HIV
Keywords: nicotine replacement therapy; antiretroviral; smartphone
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Usual Care (Placebo Comparator): Participants will receive brief advice to adhere to ART brief advice to quit smoking, 6-week supplies of nicotine-replacement therapy (NRT), and self-help materials to quit smoking and adhere to ART.
  Interventions: Drug: Nicoderm C-Q Transdermal Product; Behavioral: Adherence to Antiretroviral Therapy Counseling
- Smoking cessation only intervention (Active Comparator): Participants in this group will receive the usual care (UC) for adherence to ART, one in-person orientation sessions, 6-week supplies of NRT the "Crave-to-Quit" app, and two brief follow-up phone calls.
  Interventions: Drug: Nicoderm C-Q Transdermal Product; Behavioral: Adherence to Antiretroviral Therapy Counseling; Behavioral: Behavioral Smoking Cessation Counseling; Behavioral: "Crave-to-Quit" app
- Combined smoking cessation and HIV intervention (Experimental): Participants in this group will receive everything given in the Smoking Cessation Only arm and will also use the emocha app and will receive a tutorial explaining the app content and features. The study team will explain to participants that the app will help them in tracking dose-by-dose medication adherence by recording a video for themselves taking their medication.
  Interventions: Drug: Nicoderm C-Q Transdermal Product; Behavioral: Adherence to Antiretroviral Therapy Counseling; Behavioral: Behavioral Smoking Cessation Counseling; Behavioral: "Crave-to-Quit" app; Behavioral: vDOT "emocha" app

INTERVENTIONS:
Drug: Nicoderm C-Q Transdermal Product — 6 weeks of GlaxoSmithKline Nicoderm CQ (NRT)
  Other Names: NRT
Behavioral: Adherence to Antiretroviral Therapy Counseling — Brief counseling on adhering to antiretroviral therapy with self-help materials.
Behavioral: Behavioral Smoking Cessation Counseling — One time face-to-face smoking cessation counseling and 2 follow-up phone calls.
  Arms: Combined smoking cessation and HIV intervention; Smoking cessation only intervention
Behavioral: "Crave-to-Quit" app — Evidence-based mindfulness smoking cessation smartphone app ("Crave-to-Quit") adapted from an in-person mindfulness training relapse prevention smoking cessation intervention.
  Arms: Combined smoking cessation and HIV intervention; Smoking cessation only intervention
Behavioral: vDOT "emocha" app — Video Directly Observed Therapy (vDOT) smartphone app ("emocha") that allows participants to take a video of themselves taking medication to ensure adherence.
  Arms: Combined smoking cessation and HIV intervention

SUMMARY:
The purpose of this study is to learn if a mindfulness-based smoking cessation smartphone app can help people quit smoking and stay on antiretroviral therapies.

DETAILED DESCRIPTION:
The current study aims to test the feasibility of a three-arm randomized clinical trial testing the combined mindfulness training + Emocha apps intervention versus the mindfulness training app only with brief advice to improve ART adherence and usual care (UC; brief advice to quit and improve ART adherence). Our primary hypothesis is that the combination of mindfulness training + Emocha apps would be superior to the mindfulness training app with brief advice to improve ART adherence, and these two interventions would be superior to the UC in terms of the feasibility, acceptability, and potential efficacy (3-month smoking cessation; improvement in adherence to ART).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Diagnosed with HIV
* Have been prescribed ART medication in the prior 6 months
* Have smoked ≥ 5 cigarettes/day in the past year
* Be interested in making a quit attempt in the next 30 days
* Own a smartphone (apple/android)and plan to keep it active for the following 3 months
* Read/speak English
* Be able to provide consent
* Have no plans to move in the next 3 months
* Not pregnant or planning to be pregnant in the following 3 months

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners
* Have contraindication to NRT (past month myocardial infarction, history of serious arrhythmias/or unstable angina pectoris, dermatological disorder)
* Currently being treated for a psychiatric condition
* Currently being treated for smoking cessation, alcoholism, or illicit drug use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2020-10-14 (Actual); Study Completion 2020-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taghrid Asfar, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care | Smoking Cessation Only Intervention | Combined Smoking Cessation and HIV Intervention
Started | 13 | 13 | 13
Completed | 12 | 11 | 13
Not Completed | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Smoking Cessation Only Intervention | Combined Smoking Cessation and HIV Intervention | Total
Number analyzed (Participants) | 13 | 13 | 13 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.83 (5.49) | 52.54 (10.00) | 51.38 (10.06) | 52.55 (8.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 4 | 18
  Male | 6 | 6 | 9 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 1 | 3 | 1 | 5
  Non-Hispanic Black | 12 | 8 | 11 | 31
  Hispanic | 0 | 1 | 1 | 2
  Other | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Smoking Cessation
Description: Participants who self-report seven days of non-smoking.
Time Frame: Up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Smoking Cessation Only Intervention | Combined Smoking Cessation and HIV Intervention
Number analyzed (Participants) | 12 | 11 | 13
Participants | 3 | 5 | 7

2. Primary Outcome: Number of Participants With ≥ 95% Adherence to ART Medication Based on the Visual Analogue Scale
Description: Number of participants with ≥ 95% Adherence to ART Medication Based on the Visual Analogue Scale ranging from 0 to 100%. The ART medication visual analogue scale is an instrument for patients to rate their dose taken percentages (≥ 95% of doses taken will be regarded as good adherence). Higher score (0 to 100%) indicates higher adherence to ART.
Time Frame: 3 months
Measure: Number; unit: Participants
Arm/Group | Usual Care | Smoking Cessation Only Intervention | Combined Smoking Cessation and HIV Intervention
Number analyzed (Participants) | 12 | 11 | 13
Participants | 4 | 7 | 7

3. Primary Outcome: Usability of Intervention Questionnaire Score
Description: The usability of the Craving-to Quit and Emocha apps will be assessed via a questionnaire with scores ranging from 0-10 with the higher score indicating increased comfortability with using the app.
Time Frame: 3 months
Population: The usual care arm did not receive the Craving-to-Quit and Emocha App. The Smoking Cessation Only Arm only received the Craving-to-Quit App and not the Emocha app. The Combined Smoking Cessation and HIV arm received both the Craving-to-Quit and Emocha apps.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Smoking Cessation Only Intervention | Combined Smoking Cessation and HIV Intervention
Number analyzed (Participants) | 0 | 11 | 13
score on a scale
  Craving-to-Quit app |  | 8.70 (3.2) | 8.8 (1.6)
  Emocha app: number analyzed (Participants) | 0 | 0 | 13
  Emocha app |  |  | 4.4 (4.6)

4. Primary Outcome: Acceptability of Intervention Questionnaire Scores
Description: The acceptability is be assessed by 3 items "How satisfied were you with the intervention?", "How likely are you to recommend this intervention to a friend?" and "How useful was the intervention?" Each question is scored from 0-10 with the higher score indicating increased acceptability.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Smoking Cessation Only Intervention | Combined Smoking Cessation and HIV Intervention
Number analyzed (Participants) | 12 | 11 | 13
score on a scale
  How satisfied were you with the intervention? | 7.8 (2.1) | 9.3 (1.2) | 8.5 (1.9)
  How likely are you to recommend this intervention to a friend? | 5.6 (2.9) | 9.8 (0.6) | 9 (1.6)
  How useful was the intervention? | 7.4 (3.5) | 9.7 (0.7) | 8.6 (2.2)

5. Primary Outcome: Number of Participants Reporting Engagement With the Intervention
Description: Participant engagement is evaluated via self-reported use of the Craving-to-Quit and Emocha apps. Participants will complete a questionnaire indicating how often they used the apps. The response categories include: Everyday, often, some days, not often, not at all. We report the number of participants in each category or combination of categories.
Time Frame: Up to 3 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Smoking Cessation Only Intervention | Combined Smoking Cessation and HIV Intervention
Number analyzed (Participants) | 0 | 11 | 13
Participants
  For how many days did you use the Craving-to-Quit app?: Everyday/often |  | 6 | 7
  For how many days did you use the Craving-to-Quit app?: Some days/not often |  | 3 | 5
  For how many days did you use the Craving-to-Quit app?: Not at all/missing |  | 2 | 1
  How many days did you use the Emocha app?: number analyzed (Participants) | 0 | 0 | 13
  How many days did you use the Emocha app?: Everyday/often |  |  | 2
  How many days did you use the Emocha app?: Some days/not often |  |  | 5
  How many days did you use the Emocha app?: Not at all/missing |  |  | 6

6. Primary Outcome: Feasibility of Delivery
Description: The feasibility of delivery will be assessed via evaluating the:
  1. eligible, defined as number of participants eligible out of total screened
  2. recruitment rate, defined as number of participants enrolled out of total screened
  3. total completing all study activities, defined as the number of participants completing all activities out of total enrolled
Time Frame: At screening through study completion (up to 3 months)
Population: Total sample of participants from all 3 arms (n=39) and total screened (n=105).
Measure: Count of Participants; unit: Participants
Groups:
- All Participants Combined: Total sample of participants from all 3 arms
Arm/Group | All Participants Combined
Number analyzed (Participants) | 105
Participants
  Recruitment rate (Number of enrolled participants) | 39
  Number of participants completing all activities: number analyzed (Participants) | 39
  Number of participants completing all activities | 36

7. Secondary Outcome: Number of Participants With Reported Relapse
Description: Number of participants who have smoked at least once per week on two consecutive weeks after smoking cessation was confirmed.
Time Frame: Up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Smoking Cessation Only Intervention | Combined Smoking Cessation and HIV Intervention
Number analyzed (Participants) | 12 | 11 | 13
Participants | 10 | 7 | 7

8. Secondary Outcome: Number of Cigarettes Smoked Per Day
Description: Self-reported number of cigarettes smoked per day by each participant (Q. On average, how many cigarettes do you smoke per day?) at baseline assessment and at 3-month assessment.
Time Frame: At baseline and at 3 months
Measure: Mean (Standard Deviation); unit: number of cigarettes smoked per day
Arm/Group | Usual Care | Smoking Cessation Only Intervention | Combined Smoking Cessation and HIV Intervention
Number analyzed (Participants) | 12 | 11 | 13
number of cigarettes smoked per day
  Baseline | 11.42 (10.45) | 10.25 (8.06) | 9.18 (4.31)
  3 months | 6.82 (9.68) | 2.15 (2.21) | 2.64 (3.65)

ADVERSE EVENTS:
Time Frame: Up to 3 months
Arm/Group | Usual Care | Smoking Cessation Only Intervention | Combined Smoking Cessation and HIV Intervention
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2020-06-29): https://cdn.clinicaltrials.gov/large-docs/11/NCT03999411/Prot_001.pdf